CLINICAL TRIAL: NCT04882202
Title: Effect of Acetaminophen on the Incidence of Acute Kidney Injury in Patients Undergoing Aortic Surgery With Moderate Hypothermic Circulatory Arrest
Brief Title: Acetaminophen and AKI After Aortic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Yeon Ham, Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2021-0087
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Aortic Surgery
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen group (Experimental): patients receiving acetaminophen
  Interventions: Drug: Acetaminophen
- Placebo group (Placebo Comparator): patients receiving equal amount of normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1g IV every 6 hours for a weight > 50kg (maximum of 4g per 24 hours) or 15mg/kg every 6 hours for a weight < 50kg (maximum of 75mg/kg per 24 hours)
  Arms: Acetaminophen group
Other: Placebo — Normal saline 100 ml (equal amount of acetaminophen) IV every 6 hours
  Arms: Placebo group

SUMMARY:
Acute kidney injury is commonly accompanied major complication after aortic surgery.

Cardipulmonary bypass lyses erythrocyte and induces lipid peroxidation. This increases plasma free hemoglobin, F2-isoprostane, and isofuran concentration. Cell free hemoglobin have been reported to be associated with poor prognosis such as acute kidney injury, myocardial infarction, and death.

Acetaminophen is reported to attenuate hemeprotein mediated lipid peroxidation. Thus, investigators hypothesized that acetaminophen might have protective effect on the incidence of acute kidney injury in patients undergoing aortic surgery with moderate hypothermic circulatory arrest.

ELIGIBILITY:
Inclusion Criteria:

1) Patients undergoing aortic surgery with moderate hypothermic circulatory arrest.

Exclusion Criteria:

1. patients with chronic kidney disease or with dialysis, eGFR < 15ml/min/1.73m2
2. allergy to acetaminophen or propacetamol HCl
3. history of liver cirrhosis or total bilirubin > 2.0mg/dL

3) patients taking acetaminophen or diclofenac 4) patients who cannot understand informed consent

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury after aortic surgery with moderate hypothermic circulatory arrest | Postoperative 7 days
  Compare the incidence of acute kidney injury within 7 days after surgery. Acute kidney injury is defined using KDIGO criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson SA, Zaccagni H, Bichell DP, Christian KG, Mettler BA, Donahue BS, Roberts LJ 2nd, Pretorius M. Acetaminophen attenuates lipid peroxidation in children undergoing cardiopulmonary bypass. Pediatr Crit Care Med. 2014 Jul;15(6):503-10. doi: 10.1097/PCC.0000000000000149. PMID 24732290